CLINICAL TRIAL: NCT00234819
Title: A Double-Blind, Randomized, Placebo-Controlled, Efficacy and Safety Study of Bazedoxifene/Conjugated Estrogen Combinations for Treatment of Vasomotor Symptoms Associated With Menopause
Brief Title: Study Evaluating Bazedoxifene/Conjugated Estrogen Combinations in Symptoms Associated With Menopause
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 3115A1-305
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Vasomotor Symptoms Associated With Menopause
Keywords: Menopause
MeSH Terms: interventions — bazedoxifene; Estrogens, Conjugated (USP)

INTERVENTIONS:
Drug: Bazedoxifene/Conjugated Estrogen

SUMMARY:
The purpose of this study is to determine whether bazedoxifene/conjugated estrogens combinations are effective in the treatment of moderate to severe vasomotor symptoms associated with menopause.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, postmenopausal women, aged 40 to 64, with last natural menstrual period completed at lease 6 months ago
* Intact uterus
* Seeking treatment for hot flushes and experiencing 7 moderate to severe hot flushes per day or 50 per week

Exclusion Criteria:

* History of active presence of thrombophlebitis, thrombosis, thromboembolic disorders
* History of active presence of stroke, TIA, heart attack or ischemic heart disease
* History of melanoma, breast or any gynecologic cancer at any time; history of any other cancer within the past 5 years

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 325
Dates: Start 2005-10; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Number and severity of moderate and severe hot flashes at week 4 and at week 12, as reported daily on subject diary cards.

SECONDARY OUTCOMES:
Breast pain throughout the 12 week study, as reported daily on subject diary cards. Sleep scales and sleep quantity at week 4 and week 12, as indicated on a subject-completed questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (7):
- United States (7):
  - Phoenix, Arizona
  - Fort Myers, Florida
  - North Port Richey, Florida
  - Scarborough, Maine
  - Albuquerque, New Mexico
  - Winston-Salem, North Carolina
  - Pottstown, Pennsylvania

REFERENCES:
- [Derived] Archer DF, Freeman EW, Komm BS, Ryan KA, Yu CR, Mirkin S, Pinkerton JV. Pooled Analysis of the Effects of Conjugated Estrogens/Bazedoxifene on Vasomotor Symptoms in the Selective Estrogens, Menopause, and Response to Therapy Trials. J Womens Health (Larchmt). 2016 Nov;25(11):1102-1111. doi: 10.1089/jwh.2015.5558. Epub 2016 Sep 27. PMID 27676118